CLINICAL TRIAL: NCT02246621
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of Nonsteroidal Aromatase Inhibitors (Anastrozole or Letrozole) Plus LY2835219, a CDK4/6 Inhibitor, or Placebo in Postmenopausal Women With Hormone Receptor-Positive, HER2-Negative Locoregionally Recurrent or Metastatic Breast Cancer With No Prior Systemic Therapy in This Disease Setting
Brief Title: A Study of Nonsteroidal Aromatase Inhibitors Plus Abemaciclib (LY2835219) in Postmenopausal Women With Breast Cancer
Acronym: MONARCH 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15417; I3Y-MC-JPBM (Other: Eli Lilly and Company); 2014-001502-18 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: MONARCH 3
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Anastrozole; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abemaciclib + NSAI (Experimental): 150 milligrams (mg) Abemaciclib orally every 12 hours plus either 1 mg anastrozole or 2.5 mg letrozole orally once daily for 28 days (28 day cycles).
  Interventions: Drug: Abemaciclib; Drug: Anastrozole; Drug: Letrozole
- Placebo + NSAI (Placebo Comparator): Placebo orally every 12 hours plus either 1 mg anastrozole or 2.5 mg letrozole orally once daily for 28 days (28 day cycles).
  Interventions: Drug: Anastrozole; Drug: Letrozole; Drug: Placebo

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib + NSAI
Drug: Anastrozole — Administered orally
Drug: Letrozole — Administered orally
Drug: Placebo — Administered orally
  Arms: Placebo + NSAI

SUMMARY:
The main purpose of this study is to evaluate how effective nonsteroidal aromatase inhibitors (NSAI) plus abemaciclib are in postmenopausal women with breast cancer. Participants will be randomized to abemaciclib or placebo in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer
* Have locoregionally recurrent disease not amenable to resection or radiation therapy with curative intent or metastatic disease
* Have postmenopausal status
* Have either measurable disease or nonmeasurable bone-only disease
* Have a performance status ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have adequate organ function
* Have discontinued previous localized radiotherapy for palliative purposes or for lytic lesions at risk of fracture prior to randomization and recovered from the acute effects of therapy
* Are able to swallow capsules

Exclusion Criteria:

* Have visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis
* Have inflammatory breast cancer
* Have clinical evidence or a history of central nervous system (CNS) metastasis
* Are currently receiving or have previously received endocrine therapy for locoregionally recurrent or metastatic breast cancer
* Have received prior (neo)adjuvant endocrine therapy with a disease-free interval ≤12 months from completion of treatment
* Are currently receiving or have previously received chemotherapy for locoregionally recurrent or metastatic breast cancer
* Have received prior treatment with everolimus
* Have received prior treatment with any cyclin-dependent kinase (CDK) 4/6 inhibitor (or participated in any CDK4/6 inhibitor clinical trial for which treatment assignment is still blinded)
* Have initiated bisphosphonates or approved receptor activator of nuclear factor kappa-B ligand (RANK-L) targeted agents <7 days prior to randomization
* Are currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of randomization for a nonmyelosuppressive or myelosuppressive agent, respectively
* Have had major surgery within 14 days prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (154):
- United States (19):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - CBCC Global Research, Inc., Bakersfield, California
  - California Cancer Associates Research and Excellence, Fresno, California
  - TRIO-US (Translational Research in Oncology-US), Los Angeles, California
  - Central Coast Medical Oncology Corporation, Los Angeles, California
  - Orlando Health, Inc, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Los Angeles, California
  - UCLA Hematology/Oncology - Parkside, Santa Monica, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Candler Medical Oncology Practice - Statesboro, Savannah, Georgia
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Nebraska Hematology-Oncology, P.C., Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Mount Sinai Cancer Center, New York, New York
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Oncology Consultants P.A., Houston, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
- Australia (8):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Mater Adult Hospital Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Barwon Health - The Geelong Hospital, Geelong, Victoria
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (5):
  - Medizinische Universitaet Graz, Graz, Styria
  - Medizinische Universitaet Innsbruck, Innsbruck, Tyrol
  - Ordensklinikum Linz, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna, Vienna
- Belgium (6):
  - Iridium Kankernetwerk Wilrijk en Antwerp, Wilrijk, Antwerpen
  - Cliniques universitaires Saint-Luc, Brussels, Brussels Capital
  - Institut Jules Bordet, Anderlecht, Bruxelles-Capitale, Région de
  - Grand Hopital de Charleroi-Site Notre-Dame, Charleroi
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
  - AZ Delta, Roeselare
- Canada (8):
  - Cross Cancer Institute, Edmonton, Alberta
  - Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital (Ontario), Toronto, Ontario
  - Hopital Notre Dame, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux du Nord-de-l'Île-de-Montréal (CIUSSS NÎM) - H -T, Montreal, Quebec
  - Hopital du Saint-Sacrement, Québec
- France (10):
  - Polyclinique Bordeaux Nord, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan, Brest, Brittany Region
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Centre Hospitalier de Saint-Brieuc - Hôpital Yves Le Foll, Saint-Brieuc, Côtes-d'Armor
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-Roussillon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-Atlantique
  - Polyclinique de Gentilly, Nancy, Meurthe-et-Moselle
  - CHD Vendee, La Roche-sur-Yon, Vendée
  - CHU de Besancon Hopital Jean Minjoz, Besançon
- Germany (8):
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Rechts der Isar der TU München, München, Bavaria
  - Helios Dr. Horst Schmidt Kliniken, Wiesbaden, Hesse
  - Marien-Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Lübecker Onkologische Schwerpunktpraxis, Lübeck, Schleswig-Holstein
  - Facharztzentrum Eppendorf, Hamburg
  - Kath. Marienkrankenhaus gGmbH, Hamburg
- Alexandra Hospital, Athens, Attikí, Greece
- Israel (8):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Rambam Health Care Campus, Haifa, Ḥeifā
- Italy (11):
  - Ospedale Perrino, Brindisi, BR
  - Azienda Ospedaliero Universitaria di Ferrara, Cona, Ferrara
  - Ospedale San Martino, Genoa, Liguria
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Nuovo Ospedale di Prato-S.Stefano, Prato, Tuscany
  - Ospedale Sacro Cuore Don G. Calabria, Negrar, Verona
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Ospedale Bellaria - Azienda USL di Bologna, Bologna
  - Azienda Ospedaliera Ospedali Riuniti Papardo Piemonte, Messina
  - Policlinico Ospedale S. Andrea, Roma
  - Azienda Ospedaliera Santa Maria Terni, Terni
- Japan (19):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Chiba cancer center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kindai University Hospital- Osakasayama Campus, Ōsaka-sayama, Osaka
  - Saitama Prefectural Cancer Center, Kitaadachi-Gun, Saitama
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Met Cancer & Infectious Diseases Center Komagome Hp, Bunkyo-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hospital, Hiroshima
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Osaka Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
- Mexico (9):
  - Clinica Oncológica San Francisco, Torreón, Coahuila
  - Superare Centro de Infusion, México, Federal District
  - Fundacion Rodolfo Padilla AC, León, Guanajuato
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Hospital La Raza, Mexico City, Mexico City
  - Grupo Medico Camino Sc, Mexico City, Mexico City
  - Centro Oncologico Belenus, Cuernavaca, Morelos
  - Centro de Estudios Y Prevencion Del Cancer, Juchitán de Zaragoza, Oaxaca
  - Cancerología, Colinas Del Cimatario, Querétaro
- Netherlands (2):
  - Haga Ziekenhuis locatie Leyweg, The Hague, South Holland
  - Leids Universitair Medisch Centrum, Leiden
- Auckland City Hospital, Auckland, New Zealand
- Russia (7):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Fed State Budgetary Inst "N.N. Blokhin Med Center of Oncology" MHRF, Moscow, Moscow
  - European Medical Center, Moscow, Russian Federation
  - Clinic Complex, Saint Petersburg, Russian Federation
  - Republic Oncology Dispensary of MoH of Republic Tatarstan, Kaznan, Russia
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg
  - Rosmedtech Scientific Research Institute of Oncology, Saint Petersburg
- Slovakia (2):
  - Onkologicky Ustav sv. Alzbety, Bratislava, Bratislava Region
  - Vychodoslovensky Onkologicky ustav a.s., Košice, Košice Region
- South Korea (9):
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [Incheon]
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyungpook National University Chilgok Hospital, Daegu, Taegu-Kwangyǒkshi
  - Ulsan University Hospital, Ulsan, Ulsan-Kwangyǒkshi
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badajoz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donostia / San Sebastian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gävle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Örebro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Västerås
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beidou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhonghe
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malatya
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bebbington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Goetz MP, Toi M, Campone M, Sohn J, Paluch-Shimon S, Huober J, Park IH, Tredan O, Chen SC, Manso L, Freedman OC, Garnica Jaliffe G, Forrester T, Frenzel M, Barriga S, Smith IC, Bourayou N, Di Leo A. MONARCH 3: Abemaciclib As Initial Therapy for Advanced Breast Cancer. J Clin Oncol. 2017 Nov 10;35(32):3638-3646. doi: 10.1200/JCO.2017.75.6155. Epub 2017 Oct 2. PMID 28968163
- [Result] Johnston S, Martin M, Di Leo A, Im SA, Awada A, Forrester T, Frenzel M, Hardebeck MC, Cox J, Barriga S, Toi M, Iwata H, Goetz MP. MONARCH 3 final PFS: a randomized study of abemaciclib as initial therapy for advanced breast cancer. NPJ Breast Cancer. 2019 Jan 17;5:5. doi: 10.1038/s41523-018-0097-z. eCollection 2019. PMID 30675515
- [Derived] Hong J, Chen T, Ouyang L, Du N, Li A, Zhou Z, Zhang H, Xia Z, Meng J. Cost-effectiveness comparison of dalpiciclib and abemaciclib combined with an aromatase inhibitor as first-line treatment for HR+/HER2- advanced breast cancer. Expert Rev Pharmacoecon Outcomes Res. 2024 Apr;24(4):559-566. doi: 10.1080/14737167.2024.2330542. Epub 2024 Mar 20. PMID 38470447
- [Derived] Rugo HS, Harmer V, O'Shaughnessy J, Jhaveri K, Tolaney SM, Cardoso F, Bardia A, Maheshwari VK, Tripathi S, Haftchenary S, Pathak P, Fasching PA. Quality of life with ribociclib versus abemaciclib as first-line treatment of HR+/HER2- advanced breast cancer: a matching-adjusted indirect comparison. Ther Adv Med Oncol. 2023 Feb 24;15:17588359231152843. doi: 10.1177/17588359231152843. eCollection 2023. PMID 36861085
- [Derived] Takahashi M, Tokunaga E, Mori J, Tanizawa Y, van der Walt JS, Kawaguchi T, Goetz MP, Toi M. Japanese subgroup analysis of the phase 3 MONARCH 3 study of abemaciclib as initial therapy for patients with hormone receptor-positive, human epidermal growth factor receptor 2-negative advanced breast cancer. Breast Cancer. 2022 Jan;29(1):174-184. doi: 10.1007/s12282-021-01295-0. Epub 2021 Oct 18. PMID 34661821
- [Derived] Goetz MP, Okera M, Wildiers H, Campone M, Grischke EM, Manso L, Andre VAM, Chouaki N, San Antonio B, Toi M, Sledge GW Jr. Safety and efficacy of abemaciclib plus endocrine therapy in older patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: an age-specific subgroup analysis of MONARCH 2 and 3 trials. Breast Cancer Res Treat. 2021 Apr;186(2):417-428. doi: 10.1007/s10549-020-06029-y. Epub 2021 Jan 3. PMID 33392835
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30675515/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are participants who died.
Groups:
- Abemaciclib + NSAI (Nonsteroidal Aromatase Inhibitors): 150 milligrams (mg) Abemaciclib orally every 12 hours plus either 1 mg anastrozole or 2.5 mg letrozole orally once daily for 28 days (28 day cycles).
Period: Overall Study
Arm/Group | Abemaciclib + NSAI (Nonsteroidal Aromatase Inhibitors) | Placebo + NSAI
Started | 328 | 165
Received At Least One Dose of Study Drug | 327 | 161
Completed | 63 | 30
Not Completed | 265 | 135
Not completed — Withdrawal by Subject | 28 | 16
Not completed — Lost to Follow-up | 1 | 0
Not completed — On Study Treatment/ Follow Up | 236 | 119

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI | Total
Number analyzed (Participants) | 328 | 165 | 493
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.13 (9.92) | 62.92 (9.96) | 63.05 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 328 | 165 | 493
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 12 | 44
  Not Hispanic or Latino | 230 | 125 | 355
  Unknown or Not Reported | 66 | 28 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 103 | 45 | 148
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 186 | 102 | 288
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 28 | 11 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 9 | 6 | 15
  Austria | 10 | 3 | 13
  Belgium | 14 | 7 | 21
  Canada | 14 | 11 | 25
  Germany | 11 | 5 | 16
  Spain | 16 | 14 | 30
  France | 30 | 11 | 41
  United Kingdom | 7 | 2 | 9
  Greece | 0 | 1 | 1
  Israel | 28 | 19 | 47
  Italy | 11 | 11 | 22
  Japan | 38 | 15 | 53
  South Korea | 41 | 18 | 59
  Mexico | 22 | 7 | 29
  Netherlands | 2 | 4 | 6
  New Zealand | 1 | 0 | 1
  Russia | 13 | 6 | 19
  Slovakia | 2 | 0 | 2
  Sweden | 3 | 1 | 4
  Turkey | 9 | 3 | 12
  Taiwan | 23 | 9 | 32
  United States | 24 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time from the first day of therapy to the first evidence of disease progression as defined by RECIST v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Randomization to Progressive Disease or Death Due to Any Cause (Up to 32 Months)
Population: All randomized participants who had evaluable data. Censored participants: Abemaciclib + NSAI = 190 and Placebo + NSAI =57.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Abemaciclib + NSAI: 150 mg Abemaciclib orally every 12 hours plus either 1 mg anastrozole or 2.5 mg letrozole orally once daily for 28 days (28 day cycles).
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
Months | 28.18 [23.51 to NA] — The upper limit of the 95% CI was not evaluable due to the high censoring rate. | 14.76 [11.24 to 19.20]
Statistical Analysis 1: Comparison: Abemaciclib + NSAI vs Placebo + NSAI; Test type: Superiority; p = 0.000002, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.418 to 0.698]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from first dose date to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Time Frame: Randomization to Progressive Disease or Death Due to Any Cause (Estimated Up to 82 Months)
Reporting Status: Not Posted, anticipated posting 2026-12

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Randomization to Progressive Disease or Death Due to Any Cause (Up to 32 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
Percentage of Participants | 49.7 [44.3 to 55.1] | 37 [29.6 to 44.3]
Statistical Analysis 1: Comparison: Abemaciclib + NSAI vs Placebo + NSAI; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel

4. Secondary Outcome: Duration of Response (DoR)
Description: DOR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date.
Time Frame: CR or PR to Disease Progression or Death Due to Any Cause (Up to 32 Months)
Population: All randomized participants who had evaluable data. Censored participants: Abemaciclib + NSAI = 112 and Placebo + NSAI =28.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 163 | 61
Months | 27.39 [25.74 to NA] — The upper limit of the 95% CI was not evaluable due to the high censoring rate. | 17.46 [11.21 to 22.19]

5. Secondary Outcome: Percentage of Participants With CR, PR or Stable Disease (SD) (Disease Control Rate [DCR])
Description: DCR was the percentage of participants with a best overall response of CR, PR, or SD as per response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Randomization to Progressive Disease or Death Due to Any Cause (Up to 32 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
Percentage of Participants | 88.7 [85.3 to 92.1] | 86.7 [81.5 to 91.9]
Statistical Analysis 1: Comparison: Abemaciclib + NSAI vs Placebo + NSAI; Test type: Superiority; p = 0.501, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants With Tumor Response of SD for at Least 6 Months, PR, or CR (Clinical Benefit Rate [CBR])
Description: CBR defined as percentage of participants with best overall response of CR, PR, or SD with a duration of at least 6 months. CR, PR, or SD were defined using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. Percentage of participants = (participants with CR+PR+SD with a duration of at least 6 months / number of participants enrolled) * 100.
Time Frame: Randomization to Progressive Disease or Death Due to Any Cause (Up to 32 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
Percentage of Participants | 78.0 [73.6 to 82.5] | 71.5 [64.6 to 78.4]
Statistical Analysis 1: Comparison: Abemaciclib + NSAI vs Placebo + NSAI; Test type: Superiority; p = 0.101, Cochran-Mantel-Haenszel

7. Secondary Outcome: Change From Baseline to End of Study in Symptom Burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Functional Scale Scores
Description: EORTC QLQ-C30 v3.0 is a self-administered questionnaire with multidimensional scales that measures 5 functional domains(physical,role,cognitive,emotional, and social),global health status, and symptom scales of fatigue, pain, nausea and vomiting,dyspnea,loss of appetite,insomnia,constipation and diarrhea, and financial difficulties.Functional scale options are defined on a 7-point scale ranging from 1, "Very poor" to 7, "Excellent". A linear transformation is applied to standardize the raw scores to range between 0 and 100 with higher score indicating better functioning. For functional domains and global health status, higher scores represent a better level of functioning. Least Square(LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, Visit, Treatment*Visit and Baseline.
Time Frame: Baseline, End of Study (Up to 32 Months)
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
score on a scale
  Physical | -1.0 (0.9) | 1.7 (1.2)
  Role | -1.4 (1.1) | 2.9 (1.6)
  Emotional | 4.7 (0.9) | 4.0 (1.3)
  Cognitive | -4.0 (0.9) | -4.0 (1.3)
  Social | -0.1 (1.0) | 3.3 (1.4)

8. Secondary Outcome: Change From Baseline to End of Study in Symptom Burden on the EORTC QLQ-C30 Symptom Scale Scores
Description: EORTC QLQ-C30 v3.0 is a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, cognitive, emotional, and social), global health status, and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties. Symptom scale ranges from: 1, "Not at all"; 2, "A little"; 3, "Quite a bit"; to 4, "Very much." A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For symptoms scales, higher scores indicated greater symptom burden. Least Square(LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, Visit, Treatment*Visit and Baseline. Small changes are generally defined as at least a 3, 4 or 5 point change from baseline.
Time Frame: Baseline, End of Study (Up to 32 Months)
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
score on a scale
  Fatigue | 2.4 (1.0) | -2.6 (1.4)
  Nausea and Vomiting | 2.4 (0.6) | -0.4 (0.9)
  Pain | -4.8 (1.0) | -5.7 (1.5)
  Dyspnea | 0.9 (1.0) | -1.6 (1.4)
  Insomnia | -1.7 (1.2) | -4.1 (1.7)
  Appetite loss | 0.2 (1.1) | -3.9 (1.6)
  Constipation | -0.8 (0.9) | 1.6 (1.3)
  Diarrhea | 18.2 (1.0) | -0.5 (1.5)
  Financial difficulties | -0.7 (1.1) | -1.2 (1.6)

9. Secondary Outcome: Change From Baseline to End of Study in Symptom Burden on the EORTC QLQ-Breast23 Questionnaire
Description: The EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual functioning, sexual enjoyment, future perspective) and four symptom scales (systemic side effects, breast symptoms, arm symptoms, upset by hair loss). QLQ-BR23 questionnaire employs 4-point scales with responses from: 1, "Not at all"; 2, "A little"; 3, "Quite a bit"; to 4, "Very much". All scores are converted to a 0 to 100 scale. A higher score representing a higher ("better") level of functioning (BR23: body image, sexual functioning, future perspective), or a higher ("worse") level of symptoms. Least Square (LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, Visit, Treatment*Visit and Baseline.
Time Frame: Baseline, End of Study (Up to 32 Months)
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
score on a scale
  Body image | -4.5 (1.1) | 0.6 (1.6)
  Sexual functioning | -0.2 (0.7) | -0.1 (1.0)
  Future perspective | 12.7 (1.3) | 11.9 (1.9)
  sexual enjoyment: number analyzed (Participants) | 0 | 0
  Systemic therapy side effects | 8.15 (0.68) | 3.68 (0.98)
  Breast symptoms | -6.12 (0.64) | -6.23 (0.93)
  Arm symptoms | -1.14 (0.87) | -2.23 (1.27)
  upset by hair loss: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline to End of Study in Health Status on the EuroQuol 5-Dimension 5 Level (EuroQol-5D 5L) Index Value
Description: The EuroQol-5D (version 5L) is a brief self-administered, validated instrument consisting of 2 parts.The first part consists of 5 descriptors of current health state (mobility, self care, usual activities, pain/discomfort, and anxiety/ depression); a participant is asked to rate each state on a five level scale (no problem, slight problem, moderate problem, severe problem and extreme problem) with higher levels indicating greater severity/ impairment. Published weights are available that allow for the creation of a single summary score called the EQ-5D index that ranges from 0 to 1, with low scores representing a higher level of dysfunction and 1 as perfect health. Minimally important differences in the EQ-5D index score are 0.06 or greater in cancer patients. Least Square(LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, Visit, Treatment*Visit and Baseline.
Time Frame: Baseline, End of Study (Up to 32 Months)
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
units on a scale | 0.01 (0.01) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Abemaciclib + NSAI vs Placebo + NSAI; Test type: Superiority; p = 0.688, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.02

11. Secondary Outcome: Change From Baseline to End of Study in Health Status on the EuroQol-5D 5L Visual Analog Scale (VAS) Scores Scale
Description: The EuroQol-5D (version 5L) is a brief self-administered, validated instrument consisting of 2 parts. The second part consists of the EQ-5D general health status as measured by a visual analog scale (EQ-5D VAS). EQ-5D VAS measures the participant's self-rated health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state). Minimally important differences in the EQ-5D VAS score are 7 or greater in cancer patients. Least Square(LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, Visit, Treatment*Visit and Baseline.
Time Frame: Baseline, End of Study (Up to 32 Months)
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
Number analyzed (Participants) | 328 | 165
millimeter (mm) | 0.49 (0.78) | 1.51 (1.15)
Statistical Analysis 1: Comparison: Abemaciclib + NSAI vs Placebo + NSAI; Test type: Superiority; p = 0.466, Mixed Models Analysis; Mean Difference (Net) = -1.01, Standard Error of Mean 1.39

12. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration-Time Curve From Time 0 Hour to Infinity [AUC(0-∞)] of Abemaciclib and Its Metabolites M2 and M20
Description: Pharmacokinetics (PK): Area Under the Plasma Concentration-Time Curve From Time 0 Hour to Infinity [AUC(0-∞)] of Abemaciclib and Its Metabolites M2 and M20
Time Frame: Cycle 1 Day 1; 2 to 4 hours (h) post dose, Cycle 2 Day 1; 3 h post dose; 7 h post dose, Cycle 3 Day 1; pre dose, 3 h post dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours/milliliter (ng*h/mL)
Arm/Group | Abemaciclib + NSAI
Number analyzed (Participants) | 322
nanogram*hours/milliliter (ng*h/mL)
  Abemaciclib | 3360 (36.6)
  M2 | 1290 (75.8)
  M20 | 2300 (74.4)

13. Secondary Outcome: PK: Hepatic Clearance of Abemaciclib, and Apparent Hepatic Clearance of Its Metabolites M2 and M20
Description: PK: Hepatic Clearance of Abemaciclib, and apparent hepatic clearance of its Metabolites M2 and M20
Time Frame: as for outcome 12
Population: All randomized participants who received at least one dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour (L/h)
Arm/Group | Abemaciclib + NSAI
Number analyzed (Participants) | 322
liters/hour (L/h)
  Abemaciclib | 23.0 (26.7)
  M2 | 21.6 (50.4)
  M20 | 26.0 (46.4)

ADVERSE EVENTS:
Time Frame: Baseline Up to 32 Months
Description: Serious Adverse Events and Other Adverse Events: All participants who received at least one dose of study drug; All-Cause Mortality: All randomized participants.
Arm/Group | Abemaciclib + NSAI | Placebo + NSAI
All-Cause Mortality (participants affected / at risk) | 63/328 | 30/165
Serious Adverse Events (participants affected / at risk) | 102/327 | 27/161
Other Adverse Events (participants affected / at risk) | 322/327 | 141/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + NSAI (N=327) | Placebo + NSAI (N=161)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
General physical health deterioration (General disorders) | 2 (2) | 1 (2)
Inflammation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 13 (17) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (6) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 8 (10) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + NSAI (N=327) | Placebo + NSAI (N=161)
Anaemia (Blood and lymphatic system disorders) | 102 (328) | 13 (21)
Leukopenia (Blood and lymphatic system disorders) | 72 (293) | 4 (6)
Lymphopenia (Blood and lymphatic system disorders) | 24 (67) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 143 (625) | 3 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 41 (91) | 5 (12)
Dry eye (Eye disorders) | 17 (19) | 1 (1)
Lacrimation increased (Eye disorders) | 23 (30) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 102 (158) | 20 (24)
Constipation (Gastrointestinal disorders) | 57 (81) | 23 (29)
Diarrhoea (Gastrointestinal disorders) | 267 (984) | 52 (97)
Dyspepsia (Gastrointestinal disorders) | 26 (33) | 5 (5)
Nausea (Gastrointestinal disorders) | 135 (239) | 33 (44)
Stomatitis (Gastrointestinal disorders) | 41 (55) | 17 (25)
Vomiting (Gastrointestinal disorders) | 98 (146) | 20 (31)
Fatigue (General disorders) | 135 (255) | 54 (79)
Influenza like illness (General disorders) | 39 (54) | 15 (19)
Oedema peripheral (General disorders) | 33 (41) | 10 (11)
Pain (General disorders) | 27 (35) | 11 (14)
Pyrexia (General disorders) | 33 (40) | 16 (19)
Upper respiratory tract infection (Infections and infestations) | 33 (48) | 9 (15)
Urinary tract infection (Infections and infestations) | 34 (46) | 16 (31)
Fall (Injury, poisoning and procedural complications) | 17 (24) | 3 (3)
Alanine aminotransferase increased (Investigations) | 57 (143) | 12 (17)
Aspartate aminotransferase increased (Investigations) | 55 (119) | 12 (14)
Blood alkaline phosphatase increased (Investigations) | 19 (25) | 6 (7)
Blood creatinine increased (Investigations) | 67 (174) | 7 (8)
Weight decreased (Investigations) | 36 (65) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 86 (140) | 17 (23)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (48) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 56 (91) | 33 (50)
Back pain (Musculoskeletal and connective tissue disorders) | 52 (67) | 26 (33)
Bone pain (Musculoskeletal and connective tissue disorders) | 33 (42) | 14 (20)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 17 (27) | 6 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 34 (38) | 12 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 35 (50) | 19 (26)
Dizziness (Nervous system disorders) | 44 (57) | 18 (20)
Dysgeusia (Nervous system disorders) | 31 (37) | 5 (5)
Headache (Nervous system disorders) | 64 (102) | 26 (37)
Neuropathy (Nervous system disorders) | 35 (42) | 16 (17)
Anxiety (Psychiatric disorders) | 11 (16) | 9 (11)
Insomnia (Psychiatric disorders) | 24 (28) | 16 (17)
Breast pain (Reproductive system and breast disorders) | 14 (20) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 48 (69) | 20 (27)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 (56) | 11 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 90 (95) | 18 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 31 (39) | 4 (4)
Nail ridging (Skin and subcutaneous tissue disorders) | 17 (20) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 47 (68) | 15 (19)
Rash (Skin and subcutaneous tissue disorders) | 50 (72) | 8 (14)
Hot flush (Vascular disorders) | 33 (34) | 28 (35)
Hypertension (Vascular disorders) | 24 (46) | 10 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (5):
  • Study Protocol: JPBM Protocol (a) (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT02246621/Prot_000.pdf
  • Study Protocol: JPBM Protocol (b) (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT02246621/Prot_003.pdf
  • Study Protocol: JPBM Protocol (2014-09-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT02246621/Prot_004.pdf
  • Statistical Analysis Plan: SAP V5 Addendum (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT02246621/SAP_001.pdf
  • Statistical Analysis Plan: SAP V5 (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02246621/SAP_002.pdf